CLINICAL TRIAL: NCT04298099
Title: Ropivacaine Plasma Concentrations and Pharmacokinetics Following Erector Spinae Plane Block in the Pediatric Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Karla Elizabeth Wyatt, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-46638
Record Dates: First submitted 2020-03-03; First posted 2020-03-06 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia, Local
Keywords: Ropivacaine; Erector spinae plane block; Pediatric
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either ropivacaine 0.2% at 0.3ml/kg or ropivacaine 0.5% at 0.3ml/kg on an odd/even basis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropivacaine 0.2% at 0.3ml/kg (Active Comparator): Ropivacaine 0.2% at 0.3ml/kg
  Interventions: Drug: Ropivacaine
- Ropivacaine 0.5% at 0.3ml/kg (Active Comparator): Ropivacaine 0.5% at 0.3ml/kg
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Given the reproducible efficacy of the erector spinae plane block for thoracic procedures, this pilot study will recruit patients scheduled to undergo thoracic surgery with the adjunct of an erector spinae plane block for perioperative pain. Participants will be assigned sequentially to either ropivacaine 0.2% at 0.3ml/kg or ropivacaine 0.5% at 0.3ml/kg.
  Other Names: Naropin

SUMMARY:
The primary aim of this study is to evaluate the pharmacokinetics of serum ropivacaine concentrations following erector spinae plane peripheral nerve blocks in the pediatric population.

Secondary outcomes will assess the efficacy of the block with perioperative morphine equivalent consumption and pain scores.

DETAILED DESCRIPTION:
This pilot study will enroll patients at Texas Children's Hospital, aged 6 months to <18 years scheduled to undergo a clinically indicated thoracic surgery with the adjunct of an erector spinae plane block for perioperative pain. A single shot erector spinae plane block is commonly offered for unilateral video-assisted thoracoscopic surgery (VATS) and unilateral chest tube insertions. Following parental consent and child assent to the block, participants will be assigned sequentially to either ropivacaine 0.2% at 0.3ml/kg or ropivacaine 0.5% at 0.3ml/kg. This pilot study poses no additional risk to the patient and the thoracic surgical procedures outlined are those for which an erector spinae plane block would be offered. Furthermore, the block dosing of 0.3ml/kg volumes with ropivacaine 0.2% or 0.5% are not outside of the standard of care or accepted dosages for peripheral nerve blocks.

Venous sample serum ropivacaine levels will be collected prior to ESP block and at 30, 60, 90-minutes and 2, 4, 6 -hours from intravenous access in situ. A baseline alpha-1 acid glycoprotein (AGP) test will be collected and processed by TCH Pathology. Amide local anesthetics are predominantly protein bound to AGP. It is the unbound form that is active. While this study seeks to understand the pharmacokinetics of ropivacaine following a single shot erector spinae plane block, correlate of the AGP will simultaneously ascertain the free vs bound portion.

Samples will be analyzed for the total and free serum ropivacaine concentrations. Pain scores will be collected from nursing records starting from arrival in the Post-Anesthesia Care Unit every 4 hours (up to 12 hours after arrival in PACU). Pain will be measured using The Face, Legs, Activity, Cry, Consolability scale (FLACC), the Wong-Baker FACES Pain Rating Scale (FACES), and the Visual Analogue Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Age: 6 months - < 18 years old;
* Chest tubes or minimally invasive video assisted thoracic surgery;
* Surgery scheduled between 7AM and 5PM
* Weight greater than 4kg

Exclusion Criteria:

* Renal dysfunction;
* Liver dysfunction;
* Hypoalbuminemia;
* Allergy to local anesthetic;
* Spinal hardware or instrumentation;
* Scoliosis;
* Obesity defined as a BMI >95% percentile

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karla Wyatt, MD, MS, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walker BJ, Long JB, Sathyamoorthy M, Birstler J, Wolf C, Bosenberg AT, Flack SH, Krane EJ, Sethna NF, Suresh S, Taenzer AH, Polaner DM, Martin L, Anderson C, Sunder R, Adams T, Martin L, Pankovich M, Sawardekar A, Birmingham P, Marcelino R, Ramarmurthi RJ, Szmuk P, Ungar GK, Lozano S, Boretsky K, Jain R, Matuszczak M, Petersen TR, Dillow J, Power R, Nguyen K, Lee BH, Chan L, Pineda J, Hutchins J, Mendoza K, Spisak K, Shah A, DelPizzo K, Dong N, Yalamanchili V, Venable C, Williams CA, Chaudahari R, Ohkawa S, Usljebrka H, Bhalla T, Vanzillotta PP, Apiliogullari S, Franklin AD, Ando A, Pestieau SR, Wright C, Rosenbloom J, Anderson T; Pediatric Regional Anesthesia Network Investigators. Complications in Pediatric Regional Anesthesia: An Analysis of More than 100,000 Blocks from the Pediatric Regional Anesthesia Network. Anesthesiology. 2018 Oct;129(4):721-732. doi: 10.1097/ALN.0000000000002372. PMID 30074928
- [Background] Suresh S, De Oliveira GS Jr. Local anaesthetic dosage of peripheral nerve blocks in children: analysis of 40 121 blocks from the Pediatric Regional Anesthesia Network database. Br J Anaesth. 2018 Feb;120(2):317-322. doi: 10.1016/j.bja.2017.10.019. Epub 2017 Nov 24. PMID 29406181
- [Background] Lonnqvist PA, Ecoffey C, Bosenberg A, Suresh S, Ivani G. The European society of regional anesthesia and pain therapy and the American society of regional anesthesia and pain medicine joint committee practice advisory on controversial topics in pediatric regional anesthesia I and II: what do they tell us? Curr Opin Anaesthesiol. 2017 Oct;30(5):613-620. doi: 10.1097/ACO.0000000000000508. PMID 28786855
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] De Cassai A, Bonvicini D, Correale C, Sandei L, Tulgar S, Tonetti T. Erector spinae plane block: a systematic qualitative review. Minerva Anestesiol. 2019 Mar;85(3):308-319. doi: 10.23736/S0375-9393.18.13341-4. Epub 2019 Jan 4. PMID 30621377
- [Background] Krishna SN, Chauhan S, Bhoi D, Kaushal B, Hasija S, Sangdup T, Bisoi AK. Bilateral Erector Spinae Plane Block for Acute Post-Surgical Pain in Adult Cardiac Surgical Patients: A Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2019 Feb;33(2):368-375. doi: 10.1053/j.jvca.2018.05.050. Epub 2018 Jun 4. PMID 30055991
- [Background] Fang B, Wang Z, Huang X. Ultrasound-guided preoperative single-dose erector spinae plane block provides comparable analgesia to thoracic paravertebral block following thoracotomy: a single center randomized controlled double-blind study. Ann Transl Med. 2019 Apr;7(8):174. doi: 10.21037/atm.2019.03.53. PMID 31168455
- [Background] Munoz F, Cubillos J, Bonilla AJ, Chin KJ. Erector spinae plane block for postoperative analgesia in pediatric oncological thoracic surgery. Can J Anaesth. 2017 Aug;64(8):880-882. doi: 10.1007/s12630-017-0894-0. Epub 2017 Apr 26. No abstract available. PMID 28447318
- [Background] Richebe P, Capdevila X, Rivat C. Persistent Postsurgical Pain: Pathophysiology and Preventative Pharmacologic Considerations. Anesthesiology. 2018 Sep;129(3):590-607. doi: 10.1097/ALN.0000000000002238. PMID 29738328
- [Background] Suresh S, De Oliveira GS Jr. Blood Bupivacaine Concentrations After Transversus Abdominis Plane Block in Neonates: A Prospective Observational Study. Anesth Analg. 2016 Mar;122(3):814-817. doi: 10.1213/ANE.0000000000001088. PMID 26579846
- [Background] Suresh S, Taylor LJ, De Oliveira GS Jr. Dose effect of local anesthetics on analgesic outcomes for the transversus abdominis plane (TAP) block in children: a randomized, double-blinded, clinical trial. Paediatr Anaesth. 2015 May;25(5):506-10. doi: 10.1111/pan.12550. Epub 2014 Oct 21. PMID 25331203
- [Background] Long JB, Birmingham PK, De Oliveira GS Jr, Schaldenbrand KM, Suresh S. Transversus abdominis plane block in children: a multicenter safety analysis of 1994 cases from the PRAN (Pediatric Regional Anesthesia Network) database. Anesth Analg. 2014 Aug;119(2):395-399. doi: 10.1213/ANE.0000000000000284. PMID 24918899
- [Background] Knudsen K, Beckman Suurkula M, Blomberg S, Sjovall J, Edvardsson N. Central nervous and cardiovascular effects of i.v. infusions of ropivacaine, bupivacaine and placebo in volunteers. Br J Anaesth. 1997 May;78(5):507-14. doi: 10.1093/bja/78.5.507. PMID 9175963
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Zhang FF, Lv C, Yang LY, Wang SP, Zhang M, Guo XW. Pharmacokinetics of ropivacaine in elderly patients receiving fascia iliaca compartment block. Exp Ther Med. 2019 Oct;18(4):2648-2652. doi: 10.3892/etm.2019.7838. Epub 2019 Aug 1. PMID 31572513
- [Background] Arvidsson T, Eklund E. Determination of free concentration of ropivacaine and bupivacaine in blood plasma by ultrafiltration and coupled-column liquid chromatography. J Chromatogr B Biomed Appl. 1995 Jun 9;668(1):91-8. doi: 10.1016/0378-4347(95)00059-r. PMID 7550986
- [Background] Yasumura R, Kobayashi Y, Ochiai R. A comparison of plasma levobupivacaine concentrations following transversus abdominis plane block and rectus sheath block. Anaesthesia. 2016 May;71(5):544-9. doi: 10.1111/anae.13414. Epub 2016 Mar 4. PMID 26945692
- [Background] Berde CB, Yaster M, Meretoja O, McCann ME, Huledal G, Gustafsson U, Larsson LE. Stable plasma concentrations of unbound ropivacaine during postoperative epidural infusion for 24-72 hours in children. Eur J Anaesthesiol. 2008 May;25(5):410-7. doi: 10.1017/S0265021507003146. Epub 2008 Jan 21. PMID 18205962
- [Background] Tucker GT. Pharmacokinetics of local anaesthetics. Br J Anaesth. 1986 Jul;58(7):717-31. doi: 10.1093/bja/58.7.717. No abstract available. PMID 3524638
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled from the hospital pre-op area. The enrollment period from Dec. 2020 to January 2021. The initial subject was enrolled on Dec. 18, 2020 and the last enrolled on January 27, 2021. All subjects enrolled met the inclusion criteria and were dosed with 0.5% ropivacaine.
Pre-assignment Details: No subjects were enrolled into the Ropivicaine 0.2% at 0.3mL/kg arm.
Period: Overall Study
Arm/Group | Ropivacaine 0.2% at 0.3ml/kg | Ropivacaine 0.5% at 0.3ml/kg
Started | 0 | 4
Completed | 0 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants given the 0.2% ropivacaine dose
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine 0.2% at 0.3ml/kg | Ropivacaine 0.5% at 0.3ml/kg | Total
Number analyzed (Participants) | 0 | 4 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 4 | 4
  Between 18 and 65 years |  | 0 | 0
  >=65 years |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States |  | 4 | 4
Weight(kg) [Number; unit: kg] — Population: Participant individual weight on day of intervention.
  kg
    weight (subject 1): number analyzed (Participants) | 0 | 1 | 1
    weight (subject 1) |  | 56.2 | 56.2
    weight (subject 2): number analyzed (Participants) | 0 | 1 | 1
    weight (subject 2) |  | 22.1 | 22.1
    weight (subject 3): number analyzed (Participants) | 0 | 1 | 1
    weight (subject 3) |  | 9.6 | 9.6
    weight (subject 4): number analyzed (Participants) | 0 | 1 | 1
    weight (subject 4) |  | 53.8 | 53.8
Dose ropivacaine 0.5% at 0.3mL/kg [Number; unit: ng/mL] — Population: The dose given for each subject was administered as appropriated for weight.
  ng/mL
    Dose (Subj. 1): number analyzed (Participants) | 0 | 1 | 1
    Dose (Subj. 1) |  | 84.3 | 84.3
    Dose (Subj. 2): number analyzed (Participants) | 0 | 1 | 1
    Dose (Subj. 2) |  | 33.15 | 33.15
    Dose (Subj. 3): number analyzed (Participants) | 0 | 1 | 1
    Dose (Subj. 3) |  | 11.50 | 11.50
    Dose (Subj. 4): number analyzed (Participants) | 0 | 1 | 1
    Dose (Subj. 4) |  | 9.37 | 9.37

OUTCOME MEASURES:

1. Primary Outcome: Ropivacaine Concentrations
Description: Pharmacokinetics(PK) of free and total serum ropivacaine concentrations following erector spinae plane peripheral nerve block administration. Blood samples were drawn at the indicated time points for each subject. Laboratory assays will be completed and resulted for all subject samples collected.
Time Frame: Prior to administration and at 30, 60, 90-minutes and 2, 4, 6-hours following intravenous access in situ
Population: All participants were given a 0.5% concentration of ropivacaine at 0.3mL/kg. PK blood samples drawn from baseline( prior to administration)up to 6 hours post dose.
  Serum concentrations was were compared across time points using the non linear mixed-effects modeling(NONREM) approach. Sode/serum concentration simulations was also utilized in analysis. Data will be reported as either mean, standard deviation or median and interquartile range as appropriate.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Total Ropivacaine Concentration (ng/mL): Ropivacaine 0.5% at 0.3ml/kg
  Ropivacaine: Given the reproducible efficacy of the erector spinae plane block for thoracic procedures, this pilot study will recruit patients scheduled to undergo thoracic surgery with the adjunct of an erector spinae plane block for perioperative pain. Participants will be assigned sequentially to either ropivacaine 0.2% at 0.3ml/kg or ropivacaine 0.5% at 0.3ml/kg.
- Free Ropivacaine Concentration (ng/mL): Ropivacaine 0.5% at 3mL/kg
Arm/Group | Ropivacaine 0.2% at 0.3ml/kg | Total Ropivacaine Concentration (ng/mL) | Free Ropivacaine Concentration (ng/mL)
Number analyzed (Participants) | 0 | 4 | 4
ng/mL
  Time (Baseline/Trough) |  | 0 (0) | 0 (0)
  Time (30min post administration) |  | 1232.25 (282.20) | 850.25 (187.19)
  Time (60 min post administration) |  | 776.25 (318.57) | 518 (151.33)
  Time (90 min post administration) |  | 949.5 (100.1) | 631 (174.73)
  Time (120 min post administration) |  | 779.5 (386.24) | 468.25 (202.10)
  Time (240 min post administration) |  | 684 (425.62) | 417 (229.83)
  Time (360 min post administration) |  | 780.5 (336.5) | 509 (146)

2. Secondary Outcome: Post-anesthesia Care Unit Pain Scores Using FLACC Scale
Description: The Face, Legs, Activity, Cry, Consolability Scale (FLACC) is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2. Scores will be tracked from nursing inputs.
  There scale was utilized for one subject. The measure data was collected <2 hours post-op.
Time Frame: Every 4 hours (up to 12 hours after arrival in PACU)
Population: Scale utilized as developmentally age appropriate.
Measure: Number; unit: score on a scale
Groups:
- Post Anesthesia Care Unit (PACU) Pain Scores Using FLACC Scale: The Face, Legs, Activity, Cry, Consolability Scale (FLACC) is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2. Scores will be tracked from nursing inputs.
Arm/Group | Post Anesthesia Care Unit (PACU) Pain Scores Using FLACC Scale
Number analyzed (Participants) | 1
score on a scale | 0

3. Secondary Outcome: Post-anesthesia Care Unit Pain Scores Using FACES Pain Rating Scale
Description: The FACES Pain Rating Scale is a tool originally created for children to help them communicate their pain. Now the scale is used around the world with people ages 3 and older. The scale uses 6 faces scored 0-10 with 0 representing no pain. Each facial criteria increases by a score of 2. Scores will be tracked from nursing inputs.
  There was no data collected for this measure as this scale was not used. Subjects were assessed with a different validated Pain Scale, not data was collected using this scale.
Time Frame: Every 4 hours (up to 12 hours after arrival in PACU)
Population: Subjects pain scores were collected using a different validated pain scale.
Groups:
- Post Anesthesia Care Unit Pain Scores Using VAS: The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." A score of 0 represents no pain and 10 represents the worst the pain could be. Scores will be tracked from nursing inputs.
Arm/Group | Post Anesthesia Care Unit Pain Scores Using VAS
Number analyzed (Participants) | 0

4. Secondary Outcome: Post-anesthesia Care Unit Pain Scores Using VAS
Description: The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." A score of 0 represents no pain and 10 represents the worst the pain could be. Scores will be tracked from nursing inputs.
Time Frame: Every 4 hours (up to 12 hours after arrival in PACU)
Population: The assessment was used when developmentally age appropriate. This scale was not used in the assessment of one subject, 3 subjects were analyzed.
Measure: Number; unit: score on a scale
Groups:
- Post Anesthesia Care Unit Pain Scores Using VAS: The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." A score of 0 represents no pain. Scores will be tracked from nursing inputs.
Arm/Group | Post Anesthesia Care Unit Pain Scores Using VAS
Number analyzed (Participants) | 3
score on a scale
  Subj. 1- Numeric Pain score < 2 hours post op: number analyzed (Participants) | 1
  Subj. 1- Numeric Pain score < 2 hours post op | 5
  Subj.2- Numeric Pain score < 2 hours post-op: number analyzed (Participants) | 1
  Subj.2- Numeric Pain score < 2 hours post-op | 1.68
  Subj. 4- Numeric Pain score < 2 hours post-op: number analyzed (Participants) | 1
  Subj. 4- Numeric Pain score < 2 hours post-op | 6

5. Secondary Outcome: Morphine Equivalents
Description: Consumption of morphine per subject was collected post-operatively.
Time Frame: 12 hours
Population: Morphine milligram equivalents(MME) obtained on each participant that was administered ropivacaine dose. MME obtained post- operatively.
Measure: Number; unit: mg
Groups:
- Morphine Equivalents: Consumption of morphine post-operatively.
Arm/Group | Morphine Equivalents
Number analyzed (Participants) | 4
mg
  Subject 1 - MME: number analyzed (Participants) | 1
  Subject 1 - MME | 5
  Subject 2- MME: number analyzed (Participants) | 1
  Subject 2- MME | 1.68
  Subject 3 - MME: number analyzed (Participants) | 1
  Subject 3 - MME | 0
  Subject 4 - MME: number analyzed (Participants) | 1
  Subject 4 - MME | 6

6. Other Pre Specified Outcome: Serum Alpha Acid Glycoprotein(AAG) Level
Description: Serum alpha acid glycoprotein levels were analyzed with serum ropivacaine concentrations. No additional samples were collected for AAG levels but laboratory analysis was completed simultaneously with ropivacaine concentrations.
Time Frame: Pre-op
Population: A sample was not collected for Subject 1
Measure: Number; unit: mg/dL
Groups:
- Alpha Acid Glycoprotein: Laboratory serum levels analyzed simultaneously with ropivacaine concentrations.
Arm/Group | Alpha Acid Glycoprotein
Number analyzed (Participants) | 3
mg/dL
  Subject 2: number analyzed (Participants) | 1
  Subject 2 | 65
  Subject 3: number analyzed (Participants) | 1
  Subject 3 | 47
  Subject 4: number analyzed (Participants) | 1
  Subject 4 | 71

ADVERSE EVENTS:
Time Frame: Length of surgery plus12 hours post-op
Description: No participants were enrolled in the 0.2% Ropivacaine arm of the study.
Groups:
- Alpha Acid Glycoprotein (AAG): Ropivacaine 0.5% Concentration of ropivacaine at 0.3mL/kg One sample was not collected.
Arm/Group | Ropivacaine 0.2% at 0.3ml/kg | Ropivacaine 0.5% at 0.3ml/kg | Alpha Acid Glycoprotein (AAG)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/0 | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT04298099/Prot_001.pdf
  • Statistical Analysis Plan (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT04298099/SAP_002.pdf